CLINICAL TRIAL: NCT03012724
Title: A Prospective Multicenter Double Blind Randomized Controlled Trial to Demonstrate That the Efficacy of the H7-Coil is as Good as the Efficacy of the H1-Coil Deep Transcranial Magnetic Stimulation (DTMS) in Subjects With Major Depression Disorder (MDD)
Brief Title: Efficacy of H7-Coil DTMS Compared to H1-Coil DTMS in Subjects With Major Depression Disorder (MDD)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Brainsway (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTP-0001-01
Record Dates: First submitted 2017-01-05; First posted 2017-01-06 (Estimated); Last update posted 2020-07-15 (Actual); Status verified 2020-01

CONDITIONS: Major Depressive Disorder (MDD)
Keywords: TMS; Deep Transcranial Magnetic Stimulation; MDD; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- H1-Coil (Active Comparator): Device: Brainsway H1-Coil Deep TMS System. An FDA cleared deep transcranial magnetic stimulation device. The coil is designed to allow deeper brain stimulation in the lateral prefrontal cortex, including the anterior cingulated cortex without a significant increase of electric fields induced in superficial cortical regions.
  Interventions: Device: H1-Coil
- H7-Coil (Experimental): Device: Brainsway H7-Coil Deep TMS System. A deep transcranial magnetic stimulation device. The coil is designed to allow deeper brain stimulation in the medial prefrontal cortex, including the anterior cingulated cortex without a significant increase of electric fields induced in superficial cortical regions.
  Interventions: Device: H7-Coil

INTERVENTIONS:
Device: H7-Coil — Deep transcranial magnetic stimulation for the treatment of major dispersion disorder with the H7-Coil
  Arms: H7-Coil
Device: H1-Coil — Deep transcranial magnetic stimulation for the treatment of major depression disorder with the FDA cleared H1-Coil
  Arms: H1-Coil

SUMMARY:
The purpose of the study is to demonstrate that the efficacy and safety of deep brain rTMS, (Transcranial Magnetic Stimulation) H7-Coil treatment as add on treatment, is as good as the FDA cleared, H1-Coil, in subjects with major depressive disorder that have been previously unsuccessfully treated with antidepressant medications.

DETAILED DESCRIPTION:
This is a prospective, 6 week, double blind, randomized, controlled, multi-center trial. The study will explore the safety and efficacy of deep brain rTMS (Transcranial Magnetic Stimulation) H7-Coil treatment and demonstrate that it is as good as the FDA cleared, H1-Coil treatment as add-on for a treatment with antidepressant drugs (a bi-therapeutic treatment ) in subjects with major depressive disorder that have been previously unsuccessfully treated with antidepressant medication.

Approximately 146 subjects will be enrolled in the study. The study population consists of subjects with MDD who have failed adequate medication treatment and who are in a current depressive episode.

The patients will be of all racial, ethnic and gender categories, ranging from 22 to 68 years of age, and have HDRS-21≥20. Outpatients will be recruited from both academic and private research centers.

The study duration is 8 weeks, with a 2 week period of screening and baseline, followed by 4 weeks of 5 daily treatments and 2 weeks of biweekly treatments. Mood and mental state will be carefully monitored through standard psychological scales and assessments during the screening and baseline and throughout treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients
* Men and women 22-68 years of age
* Primary DSM-IV diagnosis of Major Depression, single or recurrent episode.
* Current depressive episode is less than 5 years duration
* The patient did not respond to at least one but not more than four antidepressant treatments in the current episode or Patients who have not completed antidepressant trials due to intolerance to therapy of 2 or more anti-depressant medications in the current episode
* Satisfactory safety screening questionnaire for transcranial magnetic stimulation
* Patients not suffering from hypo or hyper-thyroidism based on pre-study TSH level or medically stabilized
* Capable and willing to provide informed consent and able to adhere to the treatment schedule
* Patient is stable on medication for 2 month and is not expected to change medication during all study period

Exclusion Criteria:

* Individuals diagnosed by the Investigator with the following conditions (current unless otherwise stated):

  * Depression secondary to a general medical condition, or substance-induced
  * History of substance abuse or dependence within the past 6 month (except nicotine and caffeine)
  * Any psychotic disorder (lifetime), including schizoaffective disorder, or major depression with psychotic features, Bipolar disorder, Eating disorder, Obsessive compulsive disorder
  * Post-traumatic stress disorder (current or within the past year)
  * Current generalized anxiety disorder, panic disorder or social anxiety disorder
  * Presence of a personality disorder (such as antisocial, schizotypal, histrionic, borderline, narcissistic)
* Individuals with a significant neurological disorder or insult including, but not limited to:

  * Any condition likely to be associated with increased intracranial pressure
  * Space occupying brain lesion
  * Any history of seizure EXCEPT those therapeutically induced by ECT
  * History of cerebrovascular accident
  * Transient ischemic attack within two years
  * Cerebral aneurysm
  * Dementia
  * Mini Mental State Exam score of less than or equal to 24
  * Parkinson's disease
  * Huntington's chorea
  * Multiple sclerosis
  * Increased risk of seizure for any reason
  * Individuals with hearing loss
* ECT treatment within 3 months prior to the screening visit
* History of treatment with Vagus Nerve Stimulation (VNS)
* History of treatment with Deep Brain Stimulation (DBS)
* Use of any investigational drug within 4 weeks of the randomization visit
* Use of any prohibited study medication(s)
* Present suicidal risk as assessed by the investigator or significant suicide risk
* Any self-inflicted harm in the past 3 months not in the context of suicidal ideation
* Cardiac pacemakers, implanted medication pumps, intracardiac lines, or acute, unstable cardiac disease
* Intracranial implant (e.g., aneurysm clips, shunts, stimulators, cochlear implants, or electrodes) or any other metal object within or near the head, excluding the mouth, that cannot be safely removed
* Implanted neurostimulators
* History of abnormal MRI
* Known or suspected pregnancy
* If participating in psychotherapy, must have been in stable treatment for at least 3 months prior to entry into the study, with no anticipation of change in the frequency of therapeutic sessions, or the therapeutic focus over the duration of the rTMS trial
* Clinically significant laboratory abnormality, in the opinion of the Investigator based on CBC and biochemistry
* Women of childbearing potential and not using a medically accepted form of contraception when engaging in sexual intercourse
* Women: if pregnant, planning on becoming pregnant, or currently nursing

Ages: 22 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2017-03-30 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
HDRS-21 Score Change From Baseline | Week 6 post randomization
  Change from baseline in HDRS-21 scores at week 6 post-randomization in the H7 group compared to the H1 group

SECONDARY OUTCOMES:
Response Rate in HDRS-21 | Week 6 post randomization
  Percentage of patients with reduction in HDRS-21 score from baseline in the H7 group compared to the H1 group
Remission Rate | Week 6 post randomization
  Percentage of patients in remission, at week 6 post-randomization assessment

CONTACTS AND LOCATIONS:
Locations (9):
- United States (7):
  - Kadima Neuropsychiatry, La Jolla, California
  - CalNeuro Research Group, Los Angeles, California
  - Advanced Mental Health Care Inc. - Juno Beach, Juno Beach, Florida
  - Advanced Mental Health Care Inc. - Palm Beach, Palm Beach, Florida
  - Advanced Mental Health Care Inc. - Royal Palm Beach, Royal Palm Beach, Florida
  - Medical University of South Carolina, Charleston, South Carolina
  - Greenbrook TMS NeuroHealth Centers, McLean, Virginia
- Center for Addiction & Mental Health (CAMH), Toronto, Ontario, Canada
- Dr. Hadar Shalev, Beersheba, Israel

REFERENCES:
- [Derived] Zangen A, Zibman S, Tendler A, Barnea-Ygael N, Alyagon U, Blumberger DM, Grammer G, Shalev H, Gulevski T, Vapnik T, Bystritsky A, Filipcic I, Feifel D, Stein A, Deutsch F, Roth Y, George MS. Pursuing personalized medicine for depression by targeting the lateral or medial prefrontal cortex with Deep TMS. JCI Insight. 2023 Feb 22;8(4):e165271. doi: 10.1172/jci.insight.165271. PMID 36692954